CLINICAL TRIAL: NCT02780622
Title: An Open-label, Randomized 2-period Crossover Study to Investigate the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of Warfarin in Combination With Oseltamivir in Volunteers Stabilized on Warfarin Therapy
Brief Title: A Pharmacokinetics, Pharmacodynamics and Safety Study of Warfarin in Combination With Tamiflu (Oseltamivir)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: WP21272; 2007-005037-11 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-05-23 (Estimated); Results first posted 2016-09-12 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-06

CONDITIONS: Drug Therapy, Combination
MeSH Terms: interventions — Oseltamivir; Warfarin

ARMS (2):
- First Warfarin Then Warfarin and Oseltamivir (Experimental): Participants will receive warfarin (on Days 1-5) in Treatment Period 1, followed by a washout period of at least 4 days (maximum 8 days). Participants will then receive oseltamivir 75 milligram (mg) (orally twice daily on Days 1-4 and once on Day 5) and warfarin in Treatment Period 2, and attend a follow-up visit 4-12 days after the last dose in Treatment Period 2. Participants will continue receiving warfarin once daily at a prescribed usual dose throughout the study.
  Interventions: Drug: Oseltamivir; Drug: Warfarin
- First Warfarin and Oseltamivir Then Warfarin (Experimental): Participants will receive oseltamivir 75 mg (orally twice daily on Days 1-4 and once on Day 5) and warfarin in Treatment Period 1, followed by a washout period of at least 4 days (maximum 8 days). Participants will then receive warfarin (on Days 1-5) in Treatment Period 2, and attend a follow-up visit 4-12 days after the last dose in Treatment Period 2. Participants will continue receiving warfarin once daily at a prescribed usual dose throughout the study.
  Interventions: Drug: Oseltamivir; Drug: Warfarin

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir 75 mg orally, twice daily for 4 days and once on Day 5.
  Other Names: Tamiflu®
Drug: Warfarin — Warfarin once daily, at a dose determined through titration by participants' usual hematologist.

SUMMARY:
This is an open-label, randomized, 2-period crossover study, to evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of warfarin in combination with Tamiflu (oseltamivir) in participants stabilized on warfarin. Participants will be randomized to receive either their warfarin followed oseltamivir and warfarin, or by oseltamivir and warfarin followed by warfarin. The treatment periods will be separated by a washout period of at least 4 days. Participants will continue receiving warfarin once daily at a prescribed usual dose throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been receiving warfarin once daily for at least 4 weeks prior to Screening
* Participants must have regular International Normalized ratio (INR) monitoring during warfarin therapy prior to study entry, and be willing to be trained in the use of CoaguCheck devices
* INR must fall within a target range of 2.0-3.5
* Body mass index (BMI) between 18-32 kg/m^2 inclusive

Exclusion Criteria:

* An INR value between screening and Day -1 lower than 2.0 or greater than 3.5
* A change in prescribed daily warfarin dose between Screening and Day -1
* History of any coagulopathy
* Consumption of health products or supplements containing vitamin K
* Pregnant or lactating women
* Confirmed positive urine and/or blood test for drugs of abuse at Screening or Day -1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- First Warfarin Then Warfarin and Oseltamivir: Participants received warfarin (on Days 1-5) in Treatment Period 1, followed by a washout period of at least 4 days (maximum 8 days). Participants then received oseltamivir 75 milligram (mg) (orally twice daily on Days 1-4 and once on Day 5) and warfarin in Treatment Period 2, and attended a follow-up visit 4-12 days after the last dose in Treatment Period 2. Participants continued to receive warfarin once daily at a prescribed usual dose throughout the study.
- First Warfarin and Oseltamivir Then Warfarin: Participants received oseltamivir 75 mg (orally twice daily on Days 1-4 and once on Day 5) and warfarin in Treatment Period 1, followed by a washout period of at least 4 days (maximum 8 days). Participants then received warfarin (on Days 1-5) in Treatment Period 2, and attended a follow-up visit 4-12 days after the last dose in Treatment Period 2. Participants continued to receive warfarin once daily at a prescribed usual dose throughout the study.
Period: Treatment Period 1
Arm/Group | First Warfarin Then Warfarin and Oseltamivir | First Warfarin and Oseltamivir Then Warfarin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | First Warfarin Then Warfarin and Oseltamivir | First Warfarin and Oseltamivir Then Warfarin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- All Participants: Participants were randomized to 1 of 2 treatment sequences: warfarin then oseltamivir 75 mg and warfarin; or oseltamivir 75 mg and warfarin then warfarin.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Effect-time Curve Over 96 Hours (AUEC[0-96 h]) for International Normalized Ratio (INR)
Description: INR is calculated based on results of a prothrombin time (PT) test (which measures how long it takes blood to clot) and is used to monitor individuals who are being treated with the blood-thinning medication (anticoagulant) warfarin. The net AUEC(0-96 h) was calculated using the linear trapezoidal rule; this was the area under the effect-time curve and above the baseline minus the area above the curve and below the baseline during the 5-day period. An increase in INR signifies enhancement of warfarin's anticoagulant effect.
Time Frame: Pre-dose on Day 1, 24 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), and 96 hours (Day 5)
Population: All enrolled participants.
Measure: Mean (Full Range); unit: hours*ratio
Groups:
- Warfarin: Participants who received Warfarin alone at a prescribed usual dose in treatment period 1 or treatment period 2.
- Warfarin and Oseltamivir: Participants who received warfarin at a prescribed usual dose along with oseltamivir 75 mg, orally twice daily on Days 1-4 and once on Day 5 in treatment period 1 or treatment period 2.
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
hours*ratio | -2.16 [-27.6 to 78.0] | -9.06 [-93.6 to 18.0]

2. Primary Outcome: Change From Baseline in Maximum Observed Effect (Emax) of International Normalized Ratio (INR)
Description: INR is calculated based on results of a prothrombin time (PT) test (which measures how long it takes blood to clot) and is used to monitor individuals who are being treated with the blood-thinning medication (anticoagulant) warfarin. An increase in INR signifies enhancement of warfarin's anticoagulant effect.
Time Frame: Pre-dose on Day 1, 24 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), and 96 hours (Day 5)
Population: All enrolled participants.
Measure: Mean (Full Range); unit: ratio
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
ratio | 0.3 [0.0 to 2.1] | 0.1 [0.0 to 0.5]

3. Primary Outcome: Time to Reach Maximum Change From Baseline in International Normalized Ratio (INR) (Tmax)
Description: as for outcome 2
Time Frame: Pre-dose on Day 1, 24 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), and 96 hours (Day 5)
Population: All enrolled participants.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
hours | 24.00 [0.00 to 96.0] | 0.00 [0.00 to 96.00]

4. Primary Outcome: Area Under the Plasma Effect-time Curve Over 96 Hours (AUEC[0-96 h]) for Factor VII Activity
Description: Factor VIIa is a protein that causes blood to clot, and low levels in the blood can cause excessive or prolonged bleeding after an injury or surgery. The net AUEC(0-96 h) was calculated using the linear trapezoidal rule; this was the area under the effect-time curve and above the baseline minus the area above the curve and below the baseline during the 5-day period. A decrease in factor VIIa activity signifies enhancement of warfarin's anticoagulant effect. kIU/L = 1000 * international units per liter.
Time Frame: Pre-dose on Day 1, 24 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), and 96 hours (Day 5)
Population: All enrolled participants with available data.
Measure: Mean (Full Range); unit: hours*kIU/L
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 19 | 19
hours*kIU/L | 0.568 [-9.48 to 7.56] | 1.45 [-5.16 to 12.5]

5. Primary Outcome: Change From Baseline in Maximum Observed Effect (Emax) in Factor VII Activity
Description: Factor VIIa is a protein that causes blood to clot. A decrease in factor VIIa activity signifies enhancement of warfarin's anticoagulant effect. kIU/L = 1000 * international units per liter.
Time Frame: Pre-dose on Day 1, 24 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), and 96 hours (Day 5)
Population: All enrolled participants with available data.
Measure: Mean (Full Range); unit: kIU/L
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 19 | 19
kIU/L | -0.0505 [-0.21 to 0.00] | -0.0432 [-0.15 to 0.00]

6. Primary Outcome: Time to Reach Maximum Change From Baseline in Factor VII Activity (Tmax)
Description: Factor VIIa is a protein that causes blood to clot. A decrease in factor VIIa activity signifies enhancement of warfarin's anticoagulant effect.
Time Frame: Pre-dose on Day 1, 24 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), and 96 hours (Day 5)
Population: All enrolled participants with available data.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 19 | 19
hours | 96.00 [0.00 to 96.00] | 72.00 [0.00 to 96.00]

7. Primary Outcome: Change From Baseline in Plasma Concentration of Vitamin K1
Description: Vitamin K1 is required by proteins involved in blood clotting. Food interaction with warfarin can lead to decreases in Vitamin K1 in plasma. An increase in vitamin K1 signifies enhancement of warfarin's anticoagulant effect.
Time Frame: Pre-dose on Day 1 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Full Range); unit: nanogram per liter (ng/L)
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
nanogram per liter (ng/L) | 305 [-371 to 1060] | 271 [-1100 to 1310]

8. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is an active metabolite of oseltamivir.
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 1 and 5; 18 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin and Oseltamivir
Number analyzed (Participants) | 20
hours
  Oseltamivir (Single Dose: Day 1) | 0.50 [0.50 to 3.00]
  Oseltamivir Carboxylate (Single Dose: Day 1) | 4.00 [2.00 to 6.00]
  Oseltamivir (Steady State: Day 5) | 0.75 [0.50 to 3.00]
  Oseltamivir Carboxylate (Steady State: Day 5) | 4.00 [3.00 to 6.00]

9. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for R- and S- Warfarin
Time Frame: Pre-dose; 1, 2, 4, 8, 12, 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
hours
  Total (S)-warfarin | 2.00 [1.00 to 8.13] | 4.00 [0.00 to 23.92]
  Free (S)-warfarin | 14.5 [8.74 to 53.8] | 3.01 [1.00 to 8.00]
  Total (R)-warfarin | 3.00 [1.00 to 11.83] | 4.00 [1.00 to 23.92]
  Free (R)-warfarin | 4.00 [1.00 to 11.83] | 3.00 [1.00 to 11.83]

10. Secondary Outcome: Terminal Half-life (t½) for Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is an active metabolite of oseltamivir.
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 1 and 5; 18 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Warfarin and Oseltamivir
Number analyzed (Participants) | 20
hours
  Oseltamivir (Single Dose: Day 1) | 1.77 (0.686)
  Oseltamivir Carboxylate (Single Dose: Day 1) | 6.17 (2.07)
  Oseltamivir (Steady State: Day 5) | 4.00 (3.08)
  Oseltamivir Carboxylate (Steady State: Day 5) | 8.19 (1.90)

11. Secondary Outcome: Terminal Half-life (t½) for R- and S- Warfarin
Time Frame: Pre-dose; 1, 2, 4, 8, 12, 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
hours
  Total (S)-warfarin (n = 13, 11) | 45.4 (23.0) | 45.6 (11.7)
  Total (R)-warfarin (n = 12, 12) | 56.1 (26.1) | 53.6 (12.2)

12. Secondary Outcome: Oral Plasma Clearance (CL/F) for Oseltamivir
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 1 and 5; 18 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Arm/Group | Warfarin and Oseltamivir
Number analyzed (Participants) | 20
liters per hour (L/h)
  Oseltamivir (Single Dose: Day 1) | 558 (134)
  Oseltamivir (Steady State: Day 5) | 463 (104)

13. Secondary Outcome: Oral Plasma Clearance (CL/F) for R- and S- Warfarin
Time Frame: Pre-dose; 1, 2, 4, 8, 12, 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
liters per hour (L/h)
  Total (S)-warfarin | 0.198 (0.0895) | 0.208 (0.0959)
  Free (S)-warfarin | 38.5 (17) | 38.2 (15.1)
  Total (R)-warfarin | 0.139 (0.0361) | 0.145 (0.0374)
  Free (R)-warfarin | 21.7 (5.74) | 22 (5.54)

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Oseltamivir and Oseltamivir Carboxylate
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 1 and 5; 18 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Warfarin and Oseltamivir
Number analyzed (Participants) | 20
nanogram per milliliter (ng/mL)
  Oseltamivir (Single Dose: Day 1) | 88.9 (50.0)
  Oseltamivir Carboxylate (Single Dose: Day 1) | 367 (107)
  Oseltamivir (Steady State: Day 5) | 91.2 (47.2)
  Oseltamivir Carboxylate (Steady State: Day 5) | 571 (160)

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) for R- and S- Warfarin
Description: R- and S-warfarin are two molecular versions of warfarin with slightly different structures. The reported concentrations were normalized by dividing the Cmax values (nanograms per milliliter) by the individual average dose (milligrams).
Time Frame: Pre-dose; 1, 2, 4, 8, 12, 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter/milligram (ng/mL/mg)
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
Nanogram/milliliter/milligram (ng/mL/mg)
  Total (S)-warfarin | 394 (259) | 330 (197)
  Free (S)-warfarin | 1.87 (1.30) | 1.68 (1.13)
  Total (R)-warfarin | 436 (243) | 375 (96.3)
  Free (R)-warfarin | 2.70 (1.45) | 2.37 (0.604)

16. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to 24 Hours (AUC0-24h) for Oseltamivir and Oseltamivir Carboxylate
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Warfarin and Oseltamivir
Number analyzed (Participants) | 20
h*ng/mL
  Oseltamivir (Steady state: Day 5) | 176 (38.5)
  Oseltamivir Carboxylate (Steady State: Day 5) | 7180 (2550)

17. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to 24 Hours (AUC0-24h) for R- and S- Warfarin
Description: R- and S-warfarin are two molecular versions of warfarin with slightly different structures. The reported concentrations were normalized by dividing the AUC values (hours multiplied by nanograms, per milliliter) by the individual average dose (milligrams).
Time Frame: Pre-dose; 1, 2, 4, 8, 12, 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: h*ng/mL/mg
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
h*ng/mL/mg
  Total (S)-warfarin | 6770 (4500) | 6460 (4310)
  Free (S)-warfarin | 35.2 (26.1) | 33.9 (24.1)
  Total (R)-warfarin | 7790 (2480) | 7360 (1960)
  Free (R)-warfarin | 49.4 (13.4) | 48.3 (11.9)

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to 12 Hours (AUC0-12h) for Oseltamivir and Oseltamivir Carboxylate
Time Frame: Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post-dose on Day 1 and 5; 18 and 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Warfarin and Oseltamivir
Number analyzed (Participants) | 20
h*ng/mL
  Oseltamivir (Single Dose: Day 1) | 141 (38.3)
  Oseltamivir Carboxylate (Single Dose: Day 1) | 2990 (793)
  Oseltamivir (Steady State: Day 5) | 169 (36.3)
  Oseltamivir Carboxylate (Steady State: Day 5) | 5110 (1630)

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to 12 Hours (AUC0-12h) for R- and S- Warfarin
Description: as for outcome 17
Time Frame: Pre-dose; 1, 2, 4, 8, 12, 24 hours post-dose on Day 5
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: h*ng/mL/mg
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
h*ng/mL/mg
  Total (S)-warfarin | 3610 (2200) | 3380 (2100)
  Free (S)-warfarin | 18.6 (13.0) | 17.8 (12.3)
  Total (R)-warfarin | 4140 (1320) | 3870 (1020)
  Free (R)-warfarin | 25.9 (7.84) | 24.8 (6.36)

20. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to Day 26
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Warfarin | Warfarin and Oseltamivir
Number analyzed (Participants) | 20 | 20
percentage of participants | 25.0 | 25.0

ADVERSE EVENTS:
Time Frame: Five days for each treatment period (Up to Day 26)
Description: All enrolled participants.
Arm/Group | Warfarin | Warfarin and Oseltamivir
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=20) | Warfarin and Oseltamivir (N=20)
Angina pectoris (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=20) | Warfarin and Oseltamivir (N=20)
Fungal skin infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Venipuncture site swelling (General disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.